CLINICAL TRIAL: NCT05515744
Title: Study of Pregnancy And Neonatal Health (SPAN): TIMing of dElivery (TIME) Trial
Brief Title: Study of Pregnancy And Neonatal Health (SPAN)
Acronym: SPAN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Ochsner Health System (Other); University of Pennsylvania (Other); Intermountain Health Care, Inc. (Other); Duke University (Other); Inova Fairfax Hospital (Other); University of Utah (Other); University of Alabama at Birmingham (Other); University of North Carolina, Chapel Hill (Other); Technical Resources International, Inc. (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000737; 000737-CH
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes Mellitus; Delivery Timing
MeSH Terms: conditions — Diabetes, Gestational | interventions — Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Intervention Arm 1 (Experimental): Intervention Arm 1 Experimental Initiation of Delivery by induction or planned cesarean at 37 weeks 0-2 days.
  Interventions: Procedure: Childbirth
- Intervention Arm 2 (Experimental): Intervention Arm 2 Experimental Initiation of Delivery by induction or planned cesarean at 37 weeks 3-5 days.
  Interventions: Procedure: Childbirth
- Intervention Arm 3 (Experimental): Initiation of Delivery by induction or planned cesarean at 37 weeks 6 days to 38 weeks and 1 day.
  Interventions: Procedure: Childbirth
- Intervention Arm 4 (Experimental): Intervention Arm 4 Experimental Initiation of Delivery by induction or planned cesarean at 38 weeks 2-4 days.
  Interventions: Procedure: Childbirth
- Intervention Arm 5 (Experimental): Initiation of Delivery by induction or planned cesarean at 38 weeks 5 days to 39 weeks and 0 days.
  Interventions: Procedure: Childbirth
- Intervention Arm 6 (Experimental): Intervention Arm 6 Experimental Initiation of Delivery by induction or planned cesarean at 39 weeks 1-3 days.
  Interventions: Procedure: Childbirth
- Intervention Arm 7 (Experimental): Intervention Arm 7 Experimental Initiation of Delivery by induction or planned cesarean at 39 weeks 4-6 days.
  Interventions: Procedure: Childbirth

INTERVENTIONS:
Procedure: Childbirth — Induction or planned cesarean

SUMMARY:
This study will conduct a randomized trial among women with gestational diabetes (GDM). Study of Pregnancy And Neonatal health (SPAN), TIMing of dElivery (TIME) is a randomized trial that will recruit up to 3,450 pregnant women with uncontrolled GDM and randomize the timing of their delivery. Women with GDM who are approached for the trial and are found eligible but do not consent to participating in randomization for delivery will be asked to consent for chart review only (estimated additional n=3,000). The primary objective is to determine the best time to initiate delivery for GDM-complicated deliveries (defined as the time when risk of illness and death for the newborn is the lowest) between 37-39 weeks.

DETAILED DESCRIPTION:
This is a randomized clinical trial under an adaptive design nested in a larger observational study, among women who are diagnosed with uncontrolled gestational diabetes mellitus (GDM). Women from multiple clinical sites around the United States will be recruited into the study (n=3,450). Women with GDM who are approached for the trial and are found eligible but do not consent to participating to randomization for delivery will be asked to consent for chart review only (estimated additional n=3,000). The primary objective is to determine the optimal time to initiate delivery for GDM complicated deliveries (defined as the time when neonatal morbidity and perinatal mortality risk is the lowest) between 37-39 weeks (n=3,450 women). Newborn developmental and behavior outcomes, and anthropometric measures will also be assessed as secondary outcomes, as well as an exploratory analysis to investigate whether there are clinical, non-clinical or biochemical factors such as glucose measures that will further assist in refining the interval for optimizing time of GDM complicated deliveries relative to neonatal morbidity and perinatal mortality.

ELIGIBILITY:
INCLUSION CRITERIA:

Aim 3 (GDM randomized trial, TIME) inclusion criteria:

Women inclusion criteria:

1. Age ≥ 18 Years
2. Verified diagnosis of Gestational Diabetes Mellitus (GDM) with abnormal glucose levels*** or meeting other criteria for poor control, specifically any one of the following: Estimated fetal weight ≥90th percentile (LGA), Polyhydramnios, and or Demonstrate noncompliance or nonadherence as defined clinically, including missing visits, not keeping accurate log, etc.

   ***One or more elevated fasting blood glucoses OR three or more elevated post-prandial blood glucoses after receiving education about appropriate diet and lifestyle modification (e.g. physical activity)
3. Accurate gestational age as verified by ultrasound
4. Singleton gestation
5. English or Spanish speaker
6. Plans to deliver at the study site hospital
7. Ability to provide informed consent to be randomized to initiation of delivery

EXCLUSION CRITERIA:

Aim 3 (GDM randomized trial, TIME) exclusion criteria:

1. Pre-gestational diabetes*

   *will be defined as diabetes diagnosis before pregnancy OR before 13 weeks of gestation with a documented fasting plasma glucose ≥ 126 mg/dL, random plasma glucose ≥ 200 mg/dL, 2 hour post glucose ≥ 200 mg/dL during an oral glucose tolerance test (75 g glucose load), or hemoglobin A1c ≥ 6.5%.110.
2. Previous stillbirth defined as fetal demise ≥ 20 weeks of gestation
3. Self-reported history of alcohol dependency disorder and/or other drug/substance dependency in the past year
4. Teratogen exposure (e.g. cyclophosphamide, valproic acid, warfarin)
5. Known infectious diseases associated with neonatal morbidity (e.g. malaria, cytomegalovirus, rubella, toxoplasmosis, syphilis or Zika virus)
6. Genetic disorders, aneuploidy and known major fetal anomalies
7. Fetal demise
8. Pregnancies with concurrent conditions and other indications for earlier delivery will also be excluded.
9. Participation in another interventional study that influences management of labor and delivery or perinatal morbidity or mortality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Composite of Neonatal Morbidity and Perinatal Mortality | Hospital discharge
Occurrence of Antepartum, intrapartum or neonatal death (Component of primary outcome) | Antepartum pregnancy period through Newborn Discharge
Incidence of moderate or higher neonatal respiratory support within 72 hours after birth (Component of primary outcome) | Delivery through Newborn Discharge
  Including any of the following: Nasal cannula >/= 2 LPM (liters per minute), Nasal continuous positive airway pressure (NCPAP), NIPPV; (non-invasive intermittent positive pressure ventilation; Note that NIPPV is more general than Bilevel positive airway pressure (BiPAP) i.e. BiPAP is a form of NIPPV, as is non-invasive NAVA, synchronized NIPPV, non-synchronized NIPPV, some ventilators can do nasal IMV in certain situations, etc.), Mechanical ventilation, High frequency ventilation, and ECMO/ECLS (extracorporeal mechanical support/extracorporeal life support)
Occurrence of Pneumonia (Component of primary outcome) | Delivery through Newborn Discharge
  Confirmed by X-ray or positive blood culture
Occurrence of Meconium aspiration syndrome (Component of primary outcome) | Delivery through Newborn Discharge
  Respiratory distress in an infant born through meconium-stained amniotic fluid with X-ray findings consistent with meconium aspiration syndrome, and whose symptoms could not be otherwise explained
Occurrence of Sepsis (Component of primary outcome) | Delivery through Newborn Discharge
  The diagnosis of sepsis will require the presence of a clinically ill infant in whom systemic infection is suspected with a positive blood, CSF, or catheterized/suprapubic urine culture; or, in the absence of positive cultures, clinical evidence of cardiovascular collapse or an unequivocal X-ray confirming infection.
Occurrence of Neonatal encephalopathy (Component of primary outcome) | Delivery through Newborn Discharge
  Defined by Shankaran et al. 2005
Occurrence of Intracranial hemorrhage (Component of primary outcome) | Delivery through Newborn Discharge
  Intraventricular hemorrhage grades III and IV, subgaleal hematoma, subdural hematoma, or subarachnoid hematoma
Occurrence of Seizures (Component of primary outcome) | Delivery through Newborn Discharge
Occurrence of Birth trauma (Component of primary outcome) | Delivery through Newborn Discharge
  Bone fractures, brachial plexus palsy, other neurologic injury, retinal hemorrhage, or facial nerve palsy
Occurrence of Hypotension requiring pressor support (Component of primary outcome) | Delivery through Newborn Discharge
Occurrence of hypertrophic cardiomyopathy (Component of primary outcome) | Delivery through Newborn Discharge
Incidence of neonatal intensive care unit (NICU) > 1 day (24 hours) stay | Delivery through Newborn Discharge
  NICU stay > 1 day (24 hours)

SECONDARY OUTCOMES:
Incidence of respiratory support less than moderate | Delivery through Newborn Discharge
  Hood oxygen and Nasal cannula <2 LPM (liters per minute); Other than room air (No support)
Duration of any respiratory support | Delivery through Newborn Discharge
Duration of moderate respiratory support | Delivery through Newborn Discharge
Occurrence of Transient tachypnea of the newborn | Delivery through Newborn Discharge
Occurrence of Respiratory distress syndrome in Neonates | Delivery through Newborn Discharge
  Both a clinical diagnosis and whether required surfactant
Occurrence of Hypoglycemia in neonates | Delivery through Newborn Discharge
  Glucose < 35 mg/dl) and whether required IV therapy
Occurrence of Hyperbilirubinemia in Neonates | Delivery through Newborn Discharge
  Requiring phototherapy or exchange transfusion in Neonates
Occurrence of Polycythemia in Neonates | Delivery through Newborn Discharge
  Both a clinical diagnosis and whether required partial exchange transfusion
Incidence of Therapeutic hypothermia | Delivery through Newborn Discharge
  Head or body cooling
Incidence of Transfusion of blood products or blood in neonates | Delivery through Newborn Discharge
Occurrence of neonatal intensive care unit (NICU) or intermediate care unit admission | Delivery through Newborn Discharge
Duration of Neonatal hospital stay | Delivery through Newborn Discharge
  Measured in days
Birthweight | Delivery through Newborn Discharge
Incidence of small for gestational age | Delivery through Newborn Discharge
  Defined as < 10th percentile using the Duryea reference
Incidence of large for gestational age and macrosomia | Delivery through Newborn Discharge
  LGA defined as > 90th percentile using the Duryea reference and macrosomia defined as birthweight > 4500 g
Composite of Maternal Morbidity and Mortality | Pregnancy through Discharge
  Maternal death, HELLP syndrome, Eclampsia, Pulmonary edema, placental abruption, blood transfusion
Occurrence of maternal death | Pregnancy through Discharge
Occurrence of HELLP syndrome | Pregnancy through Discharge
  As defined by American College of Obstetricians and Gynecologists (ACOG)
Occurrence of Eclampsia | Pregnancy through Discharge
  As defined by American College of Obstetricians and Gynecologists (ACOG)
Occurrence of Maternal Pulmonary edema | Pregnancy through Discharge
  Chest x-ray confirmed
Occurrence of Placental abruption | Pregnancy through Delivery
Incidence of Maternal Blood transfusion | Pregnancy through Discharge
Incidence of spontaneous labor | Pregnancy through Delivery
Incidence of induced labor | Pregnancy through Delivery
Incidence of planned cesarean | Pregnancy through Delivery
Indication for delivery including cesarean for suspected macrosomia | Pregnancy through Delivery
  Defined as estimated fetal weight > 4500 grams
Occurrence of Spontaneous vaginal delivery | Pregnancy through Delivery
Occurrence of Operative vaginal delivery | Pregnancy through Delivery
  Vacuum or forceps
Occurrence of Cesarean delivery | Pregnancy through Delivery
Indications for operative vaginal delivery | Pregnancy through Delivery
Indication for cesarean | Pregnancy through Delivery
Incidence of Shoulder dystocia | Delivery through Newborn Discharge
Occurrence of Maternal lacerations | Delivery through Discharge
  1st, 2nd, 3rd or 4th degree perineal; sulcus, vaginal wall; labial, periurethral, clitoral, abrasion, other
Occurrence of Postpartum hemorrhage | Delivery through Discharge
  Defined as any of the following: Transfusion, Non-elective hysterectomy, Use of two or more uterotonics other than oxytocin, Other surgical interventions such as uterine compression sutures, uterine artery ligation, embolization, hypogastric ligation, or balloon tamponade, and Curettage
Occurrence of Maternal ICU Admission | Delivery through Discharge
Incidence of Maternal venous thromboembolism | Delivery through Discharge
  Deep venous thrombosis or pulmonary embolism
Incidence of Chorioamnionitis | Delivery through Discharge
  Defined as a clinical diagnosis before delivery
Maternal postpartum infection | Delivery through Discharge
  Defined as, Clinical diagnosis of endometritis, Wound reopened for hematoma, seroma, infection or other reasons, Cellulitis requiring antibiotics, Pneumonia, Pyelonephritis, Bacteremia unknown source, and Septic pelvic thrombosis
Maternal hypertension | Delivery through Discharge
  Mild and Severe (systolic and diastolic) defined by ACOG
Incidence of Preeclampsia, with or without severe features | Delivery through Discharge
  Defined by ACOG
Use of antihypertensive drugs | Delivery through Discharge
  Includes oral antihypertensive, intravenous antihypertensive, or intravenous anticonvulsant
Number of hours in labor and delivery unit | Delivery through Discharge
Duration of maternal hospital stay | Pregnancy through Newborn Discharge
  Measured in Days.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Grantz, MD, MS, Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ochsner Baptist, New Orleans, Louisiana
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University Perinatal Research Center, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Intermountain Healthcare, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - INOVA Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized phenotypic data and the SNP genotype, DNA methylation, and RNA sequence data generated from the study will be deposited into scientific databases that are maintained by the National Institutes of Health.
Supporting Information: Study Protocol
Time Frame: Data will be shared before publication or at the time of publication or shortly thereafter.
Access Criteria: Access to the anonymised information stored in NIH archives like DASH and dbGaP will only be accepted via applications from appropriately qualified researchers who sign a legally-binding Data Access Agreement in which they commit to use the data only for research purposes; protect the data confidentiality; provide appropriate data security; not attempt to identify individual participants from whom data were obtained; and not redistribute the data or any subset or derivative that could be used to identify the research participant.
URL: https://dash.nichd.nih.gov/